CLINICAL TRIAL: NCT00445874
Title: A Multi-Center, Randomized, Double-Masked, Placebo-Controlled Evaluation of the Efficacy and Safety of an Anti-Allergy Drug With a Contact Lens as Compared to Placebo in the Prevention of Allergic Conjunctivitis in a Population of Allergic Contact Lens Wearers
Brief Title: Evaluation of Efficacy and Safety of an Anti-Allergy Drug With a Contact Lens in the Treatment of Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vistakon Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 06-003-23
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Allergic Conjunctivitis
Keywords: allergic conjunctivitis, ophthalmology, multicenter, controlled
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Ketotifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ketotifen with a Contact Lens (no generic name)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of an anti-allergy drug with a contact lens compared to placebo in preventing ocular itching associated with allergic conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* History of ocular allergies and a positive skin test reaction to cat hair, cat dander, grasses, ragweed, and/or trees withing the past 24 months
* Successful soft contact lens wearer who has frequently worn contact lenses for at least one month or more

Exclusion Criteria:

* Active ocular infection
* Clinically significant blepharitis
* Follicular conjunctivitis
* Pterygium
* Narrow angle glaucoma
* Dry eye dyndrome
* Ocular surgery within past 6 months
* Pregnancy or lactation

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-02; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Ocular itching

SECONDARY OUTCOMES:
Conjunctival, ciliary, and episcieral redness; chemosis and mucous discharge; tearing and lid swelling

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pall, OD, MS, FAAO, Study Director — Vistakon Pharmaceutical
Locations (6):
- United States (6):
  - Phoenix, Arizona
  - Irvine, California
  - North Andover, Massachusetts
  - Cincinnati, Ohio
  - Fairfield, Ohio
  - Mason, Ohio